CLINICAL TRIAL: NCT06648993
Title: Investigation of the Relationship Between Body Awareness and Physical Activity Levels of Pregnant Women and Age, Number of Pregnancies and Gestational Week
Brief Title: Body Awareness and Physical Activity Levels of Pregnant Women and Age, Number of Pregnancies and Gestational Week
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Aslıhan Turan, principle invastigator, KTO Karatay University
Other Study IDs: KaratayUA2
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the relationship between body awareness and physical activity levels of pregnant women according to variables such as age, number of pregnancies and gestational week. The main question it aims to answer is: do physical activity levels of pregnant women and age, number of pregnancies and gestational week have an impact on body awareness in pregnant women

ELIGIBILITY:
Inclusion Criteria:

* being in the 2-3rd trimester of pregnancy and
* volunteering to participate in the study

Exclusion Criteria:

* having a risky pregnancy,
* being prohibited from physical activity by a physician,
* having any limb deficiency,
* neurological disease,
* mental deficiency

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Body Awareness | Baseline
  The Body Awareness Questionnaire will be used to assess body awareness. The questionnaire consists of 18 questions. Participants will be asked to rate each statement on a scale ranging from 1 (1: Not true at all) to 7 (7: Completely true) and the total score will be obtained by summing the scores given for each statement. The total score takes a value between 18 and 126. The higher the total score, the better the body awareness

SECONDARY OUTCOMES:
Physical Activity Levels | Baseline
  The physical activity levels of individuals will be assessed with the International Physical Activity Questionnaire Short form (IPAQ-SF), which consists of seven questions that provide information about the number of days in the last week that the individual has engaged in high, moderate and low intensity activities, the time spent in these activities and the time spent sedentary. One criterion in this assessment is that each activity must be performed for at least 10 minutes to be included in the scoring. Minutes and days are multiplied by the metabolic equivalent of the task (MET) value and the result is expressed as MET-minutes/week. A lower value indicates a lower level of physical activity.
Age | Baseline
  Participants' age will be recorded.
Number of births | Baseline
  Participants' number of births will be recorded.
weeks of gestation | Baselin
  Participants' weeks of gestation will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)